CLINICAL TRIAL: NCT00112580
Title: Phase II Trial of Single Agent Ipilimumab (MDX-010 Anti CTLA-4) for Subjects With Locally Advanced or Metastatic Pancreatic Adenocarcinoma
Brief Title: MDX-010 in Treating Patients With Stage IV Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000430666; NCI-05-C-0141; NCI-P6557; MDX-010-24; NCT00108888 (obsolete NCT alias)
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Results first posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ipilimumab

INTERVENTIONS:
Biological: ipilimumab

SUMMARY:
RATIONALE: Biological therapies, such as MDX-010, may stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase II trial is studying how well MDX-010 works in treating patients with stage IV pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine clinical response (partial and complete responses) in patients with unresectable stage IV (locally or distantly metastatic) pancreatic adenocarcinoma treated with anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010).

Secondary

* Determine whether observed responses correlate with the incidence of autoimmunity in patients treated with this drug.

OUTLINE: This is an open-label study. Patients are stratified according to status of disease (locally vs distantly metastatic).

Patients receive anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) IV over 90 minutes on days 0, 21, 42, and 63. Treatment repeats every 84 days for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients with disease progression after achieving a partial response or complete response receive 2 additional courses of therapy.

After completion of study treatment, patients are followed at 3 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 42-82 patients (21-41 per stratum) will be accrued for this study within 2-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed pancreatic adenocarcinoma

  * Stage IV disease

    * Locally (invasion of adjacent structures, including mesenteric arteries or organs) or distantly metastatic disease
  * Unresectable disease
  * Pancreatic adenocarcinoma with intraductal papillary mucinous neoplasm allowed
* The following diagnoses are not allowed:

  * Acinar cell carcinoma
  * Pancreaticoblastoma
  * Malignant cystic neoplasms
  * Endocrine neoplasms
  * Squamous cell carcinoma
  * Vater and periampullary duodenal or common bile duct malignancies
* Clinically evaluable disease with ≥ 1 site of measurable disease
* Biliary or gastric outlet obstruction allowed provided it is effectively drained by endoscopic, operative, or interventional means
* Pancreatic, biliary, or enteric fistulae allowed provided they are controlled with an appropriate drain

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* WBC ≥ 2,500/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Hematocrit ≥ 27%

Hepatic

* Hepatitis B surface antigen negative
* Hepatitis C virus antibody negative OR
* Hepatitis C RNA negative by polymerase chain reaction

Renal

* Creatinine < 2.0 mg/dL

Immunologic

* HIV negative
* No history of or active autoimmune disease, including uveitis or autoimmune inflammatory eye disease
* No active uncontrolled infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* No underlying medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010)

Chemotherapy

* At least 3 weeks since prior chemotherapy for pancreatic adenocarcinoma and recovered
* No concurrent chemotherapy

Endocrine therapy

* More than 4 weeks since prior corticosteroids
* No concurrent systemic or topical corticosteroids

Radiotherapy

* At least 3 weeks since prior radiotherapy for pancreatic adenocarcinoma and recovered

Surgery

* See Disease Characteristics

Other

* At least 3 weeks since other prior therapy for pancreatic adenocarcinoma and recovered
* No concurrent immunosuppressants (e.g., cyclosporin or its analog)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-07-31 (Actual); Primary Completion 2009-06-30 (Actual); Study Completion 2009-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland

REFERENCES:
- [Result] Royal RE, Levy C, Turner K, Mathur A, Hughes M, Kammula US, Sherry RM, Topalian SL, Yang JC, Lowy I, Rosenberg SA. Phase 2 trial of single agent Ipilimumab (anti-CTLA-4) for locally advanced or metastatic pancreatic adenocarcinoma. J Immunother. 2010 Oct;33(8):828-33. doi: 10.1097/CJI.0b013e3181eec14c. PMID 20842054

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants were treated.
Groups:
- Locally Advanced Cohort: Participants with locally advanced pancreatic adenocarcinoma. Treated with Ipilimumab administered at 3 mg/Kg dose every 3 weeks.
- Metastatic Cohort: Participants with metastatic pancreatic adenocarcinoma. Treated with Ipilimumab administered at 3 mg/Kg dose every 3 weeks.
Period: Overall Study
Arm/Group | Locally Advanced Cohort | Metastatic Cohort
Started | 8 | 19
Completed | 0 | 0
Not Completed | 8 | 19
Not completed — Adverse Event | 1 | 2
Not completed — Disease progression | 5 | 16
Not completed — Participant withdrew consent | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Locally Advanced Cohort | Metastatic Cohort | Total
Number analyzed (Participants) | 8 | 19 | 27
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (6.48) | 51.5 (9.81) | 53.5 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 3 | 12 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 18 | 26
  Hispanic | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR)
Description: Percentage of participants who achieved Complete Response (CR) or Partial Response (PR) according to RECIST criteria. Particularly, CR is defined as disappearance of all target lesions, while PR is defined as at least a 30% decrease n the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: From first dose to 3 weeks following the end of the treatment cycle, up to 24 weeks.
Population: All treated participants
Measure: Number; unit: Percent of Participants
Arm/Group | Locally Advanced Cohort | Metastatic Cohort
Number analyzed (Participants) | 8 | 19
Percent of Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events were collected from first dose to study completion (up to approximately 1 year)
Description: Adverse Events were not monitored/assessed by disease status separately because both cohorts (Locally Advanced cohort and Metastatic cohort) received the same treatment at the same dose. Hence, Adverse Events are reported as a single cohort (Ipilimumab 3 mg/Kg).
Groups:
- Ipilimumab 3 mg/Kg: Participants with locally advanced or metastatic pancreatic adenocarcinoma treated with Ipilimumab administered at 3 mg/Kg dose every 3 weeks.
Arm/Group | Ipilimumab 3 mg/Kg
All-Cause Mortality (participants affected / at risk) | 12/27
Serious Adverse Events (participants affected / at risk) | 20/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab 3 mg/Kg (N=27)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Hypophysitis (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Jejunal ulcer (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 4
Cholangitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Liver disorder (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 2
Blood amylase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lipase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab 3 mg/Kg (N=27)
Lymphopenia (Blood and lymphatic system disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 6
Ascites (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 4
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 4
Chills (General disorders) | 4
Fatigue (General disorders) | 13
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 11
Hyperbilirubinaemia (Hepatobiliary disorders) | 5
Oral candidiasis (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 6
Haemoglobin decreased (Investigations) | 3
Weight decreased (Investigations) | 14
Weight increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2005-03-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT00112580/Prot_000.pdf
  • Statistical Analysis Plan (2009-01-06): https://cdn.clinicaltrials.gov/large-docs/80/NCT00112580/SAP_001.pdf